CLINICAL TRIAL: NCT02455869
Title: Comparative Evaluation of Subgingivally Delivered 1% Alendronate Versus 1.2% Atorvastatin Gel in Treatment of Chronic Periodontitis: a Randomized Placebo Controlled Clinical Trial
Brief Title: Comparison of Alendronate With Atorvastatin in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014J
Record Dates: First submitted 2015-05-19; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Atorvastatin; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): SRP plus placebo SRP was done for all the subjects. Placebo gel was delivered subgingivally into the pocket
  Interventions: Drug: SRP and Placebo gel
- Atorvastatin group (Active Comparator): SRP plus Atorvastatin SRP was done for all the subjects. Atorvastatin was delivered in the pocket subgingivally
  Interventions: Drug: SRP and Atorvastatin
- Alendronate Group (Active Comparator): Alendronate SRP plus Alendronate SRP was done for all the subjects. Alendronate was delivered in the pocket subgingivally
  Interventions: Drug: SRP and Alendronate

INTERVENTIONS:
Drug: SRP and Placebo gel — After SRP, placebo gel was delivered subgingivally into the pocket
  Arms: Placebo group
Drug: SRP and Atorvastatin — After SRP, Atorvastatin gel was delivered subgingivally into the pocket
  Arms: Atorvastatin group
Drug: SRP and Alendronate — After SRP, Alendronate gel was delivered subgingivally into the pocket
  Arms: Alendronate Group

SUMMARY:
The present study is designed as a single-centre, randomized, controlled clinical trial to evaluate and compare the clinical efficacy of two local drug delivery systems containing 1% ALN gel and 1.2% ATV gel in treatment of intrabony defects in patients with chronic periodontitis as an adjunct to SRP.

DETAILED DESCRIPTION:
Background: Alendronate and Atorvastatin are known to inhibit osteoclastic bone resorption and were proposed to have osteostimulative properties by causing osteoblast differentiation in vivo and in vitro as shown by an increase in matrix formation. The aim of the present study is to evaluate and compare the efficacy of 1% ALN and 1.2% ATV gel as a local drug delivery system in adjunct to scaling and root planning (SRP) for the treatment of intrabony defects in patients with chronic periodontitis.

Methods: A total of 90 intrabony defects were treated with either1%ALN, 1.2% ATV or placebo gel. Clinical parameters (plaque index, modified sulcus bleeding index, probing depth [PD], and clinical attachment level [CAL]) were recorded at baseline, 3, 6 and 9 months. Radiographic parameters intrabony defect depth (IBD) and defect depth reduction (DDR%) was calculated on standardized radiographs by using image analysis software at 6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with PDs ≥5mm or CALs ≥4 to 6mm and vertical bone loss ≥3 mm on intraoral periapical radiographs with no history of periodontal therapy or use of antibiotics in the preceding 6 months were included

Exclusion Criteria:

* Patients with a known systemic disease;
* known or suspected allergy to the ALN/bisphosphonate group and ATV/statin group;
* on systemic ALN/bisphosphonate and therapy ATV/statin group;
* with aggressive periodontitis;
* who used tobacco in any form;
* alcoholics;
* immunocompromised patients;
* and pregnant or lactating females were excluded from the study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in defect depth reduction from baseline to 6 months and from baseline to 9 months | Baseline to 6 months and Baseline to 9 months
  Radiographic defect depth reduction to measured at baseline, 6 and 9 months interval

SECONDARY OUTCOMES:
Plaque index | 3,6 and 9 months
  Plaque index will be measured at 3, 6 and 9 months
Modified sulcus bleeding index | 3,6 and 9 months]
  Modified sulcus bleeding index will be measured at 3, 6 and 9 months
Probing pocket depth | 3,6 and 9 months]
  Probing pocket depth will be measured at 3, 6 and 9 months
Clinical attachment level | 3,6 and 9 months]
  Clinical attachment level will be measured at 3, 6 and 9 months